CLINICAL TRIAL: NCT00753454
Title: A Phase IIIb, Multi-center Open-label, Follow-up Study to Evaluate the Safety and Efficacy of Certolizumab Pegol Administered Concomitantly With Methotrexate in Patients With Active Rheumatoid Arthritis Who Participated in C87077.
Brief Title: Open Label Extension for Patients Coming From the Dosing Flexibility Study in Patients With Rheumatoid Arthritis (RA)
Acronym: Dose Flex II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C87084; 2007-005267-10 (EudraCT Number)
Expanded Access: NCT03559686 (Available)
Record Dates: First submitted 2008-06-05; First posted 2008-09-16 (Estimated); Results first posted 2012-06-14 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2012-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Joint Disease; Arthritis; Certolizumab pegol; Cimzia
MeSH Terms: conditions — Arthritis, Rheumatoid; Joint Diseases; Arthritis | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CDP870 (Experimental): Patients having completed the week 34 assessment in C87077 (NCT00580840) or patients having been randomized at Week 18 and having met the pre-defined criteria for flare, will be given the option to enroll in C87084 and receive: 400 mg CZP at Entry, Week 2, and Week 4 followed by 200 mg every two weeks in combination with MTX until the drug is commercially available for the indication of RA in the patient's country or region (or until further notice from UCB).
  Interventions: Drug: Certolizumab pegol

INTERVENTIONS:
Drug: Certolizumab pegol — Liquid certolizumab pegol administered every two weeks as a single injection (400 mg at Entry, Week 2 & Week 4, followed by 200 mg every 2 weeks).
  Other Names: Cimzia

SUMMARY:
The purpose of this study is to continue to assess the safety of certolizumab pegol in combination with methotrexate (MTX).

DETAILED DESCRIPTION:
Patients having completed the week 34 assessment in the C87077 (NCT00580840) study or having met the pre-defined criteria for flare (defined as patients that have randomized at Week 18 and experienced at 2 consecutive visits between Week 18 and Week 34 inclusive an equal to Baseline (W0) or worst swollen and tender joints counts), will be given the option to enroll in C87084 and receive certolizumab pegol [400 mg at Entry, Week 2, and Week 4 followed by 200 mg every two weeks (Q2W)] in combination with MTX until the drug is commercially available for the indication of Rheumatoid Arthritis (RA) in the patient's country or region or until further notice from UCB.

All patients will continue their MTX treatment at the same stable dose as during the C87077 (NCT00580840) study, unless there is a need to reduce the dose for reasons for toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to understand the written Informed Consent Form (ICF)
* Patients must have achieved an ACR20 (American College of Rheumatology) response at Week 16 and completed the entire C87077 (NCT00580840) study or patients having been randomized at Week 18 and having met the pre-defined criteria for flare
* Patients must have complied with the protocol requirements during their participation in C87077 (NCT00580840)
* Female patients of childbearing potential must have a negative urine pregnancy test at Entry and must continue to have negative urine pregnancy tests throughout their study participation
* Patients must be willing to comply with protocol

Exclusion Criteria:

* Patients must not have a diagnosis of any other inflammatory Arthritis
* Patients must not have a secondary, non-inflammatory type of Arthritis that in the investigator's opinion is symptomatic enough to interfere with the evaluation of the study drug on the patient's primary diagnosis of Rheumatoid Arthritis (RA)
* Patients must not have a history of an infected joint prosthesis with that prosthesis still in situ
* Patients who do not meet the Medical History Exclusion criteria, as defined per protocol. Examples of exclusionary criteria (not all-inclusive): pregnancy, chronic infection, active Tuberculosis (TB), high risk of infection, Lymphproliferative Disorder, acute or chronic Viral Hepatitis B or C, known Human Immunodeficiency Virus (HIV), Malignancy or history of Malignancy, history of severe, progressive, and/or uncontrolled Renal, Hepatic, Hematological, Gastrointestinal, Endocrine, Pulmonary, Cardiac, Neurological or Cerebral Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2008-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (40):
- United States (36):
  - Huntsville, Alabama
  - Paradise Valley, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Huntington Beach, California
  - La Jolla, California
  - Los Angeles, California
  - Palm Desert, California
  - San Diego, California
  - Aventura, Florida
  - Clearwater, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - Jupiter, Florida
  - Melbourne, Florida
  - Sarasota, Florida
  - Morton Grove, Illinois
  - Vernon Hills, Illinois
  - Lexington, Kentucky
  - Haverhill, Massachusetts
  - Worcester, Massachusetts
  - Rochester, Minnesota
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - Reno, Nevada
  - Albany, New York
  - Mineola, New York
  - Syracuse, New York
  - Charlotte, North Carolina
  - Monroe, North Carolina
  - Wilmington, North Carolina
  - Norman, Oklahoma
  - Duncansville, Pennsylvania
  - Dallas, Texas
  - San Antonio, Texas
  - Tyler, Texas
- Canada (4):
  - Winnipeg, Manitoba
  - St. John's, Newfoundland and Labrador
  - St. Catharines, Ontario
  - Toronto, Ontario

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started in September 2008 with subjects from Canada and the United States. The primary completion date occurred in May 2011, with study completion in May 2011.
Pre-assignment Details: Participant Flow and Baseline Characteristics refer to the Full Analysis Set (FAS). The Full Analysis Set (FAS) consists of all subjects who were dispensed medication.
  One subject was discontinued at the discretion of investigator due to "missed visits."
Groups:
- CDP870: Patients having completed the Week 34 assessment in C87077 (NCT00580840) or patients having been randomized at Week 18 and having met the pre-defined criteria for flare, will be given the option to enroll in C87084 and receive: 400 mg CZP at Entry, Week 2, and Week 4 followed by 200 mg every two weeks in combination with MTX until the drug is commercially available for the indication of Rheumatoid Arthritis (RA) in the patient's country or region (or until further notice from UCB).
Period: Overall Study
Arm/Group | CDP870
Started | 168
Completed | 154
Not Completed | 14
Not completed — Adverse Event | 4
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 5
Not completed — Investigator Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | CDP870
Number analyzed (Participants) | 168
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 135
  >=65 years | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128
  Male | 40
Region of Enrollment [Number; unit: participants]
  United States | 157
  Canada | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Reporting At Least One Treatment-emergent Adverse Event (TEAE) During The Study Period
Description: A TEAE is defined as any untoward medical occurrence (eg, noxious or pathological changes) in a subject or clinical investigation subject compared with pre-existing conditions, that occurs during any phase of a clinical trial including Pretreatment, Run-In, Wash-Out, or Follow-Up Phases.
  A TEAE is defined as being independent of assumption of any causality (eg, to trial or concomitant medication, primary or concomitant disease, or trial design).
  TEAEs are all AEs in which the onset date and time is after the first study drug administration in C87084, up to 84 days after the last injection.
Time Frame: From Entry Visit up to approximately 60 weeks
Population: Of the 168 subjects in the Full Analysis Set (FAS), 168 are included in this analysis.
Measure: Number; unit: percentage of subjects
Arm/Group | CDP870
Number analyzed (Participants) | 168
percentage of subjects | 52.4

2. Primary Outcome: Percentage of Subjects Withdrawing From Study Due To A Treatment-emergent Adverse Event (TEAE) During The Study Period
Description: as for outcome 1
Time Frame: From Entry Visit up to approximately 60 weeks
Population: Of the 168 subjects in the Full Analysis Set (FAS), 168 are included in this analysis.
Measure: Number; unit: percentage of subjects
Arm/Group | CDP870
Number analyzed (Participants) | 168
percentage of subjects | 2.4

3. Primary Outcome: Percentage of Subjects With At Least One Treatment-emergent Serious Adverse Event (SAE) During The Study Period
Description: A Serious Adverse Event is any untoward medical occurrence that at any dose
  * results in death,
  * is life threatening,
  * requires in-patient hospitalization or prolongation of existing hospitalization,
  * results in persistent or significant disability/incapacity
  * is a congenital anomaly/birth defect
Time Frame: From Entry Visit up to approximately 60 weeks
Population: Of the 168 subjects in the Full Analysis Set (FAS), 168 are included in this analysis.
Measure: Number; unit: percentage of subjects
Arm/Group | CDP870
Number analyzed (Participants) | 168
percentage of subjects | 3.0

4. Secondary Outcome: Percentage of Subjects With ACR20 (American College of Rheumatology 20% Improvement) Response at Completion/Withdrawal Visit
Description: ACR20 response is defined for subjects with at least 20% improvement from Baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: 1) Health Assessment Questionnaire-Disability Index (HAQ-DI), 2) C-reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale, 4) Patient's Global Assessment of Disease Activity, 5) Physician's Global Assessment of Disease Activity.
Time Frame: Baseline (in C87077 [NCT00580840]) to Completion/Withdrawal Visit (up to approximately 54 weeks)
Population: Of the 168 subjects in the Full Analysis Set (FAS), 155 are included in this analysis.
  Data was not available for 13 subjects.
Measure: Number; unit: percentage of subjects
Arm/Group | CDP870
Number analyzed (Participants) | 155
percentage of subjects | 73.5

5. Secondary Outcome: Percentage of Subjects With ACR50 (American College of Rheumatology 50% Improvement) Response at Completion/Withdrawal Visit
Description: ACR50 response is defined for subjects with at least 50% improvement from Baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: 1) Health Assessment Questionnaire-Disability Index (HAQ-DI), 2) C-reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale, 4) Patient's Global Assessment of Disease Activity, 5) Physician's Global Assessment of Disease Activity.
Time Frame: Baseline (in C87077 [NCT00580840]) to Completion/Withdrawal Visit (up to approximately 54 weeks)
Population: as for outcome 4
Measure: Number; unit: percentage of subjects
Arm/Group | CDP870
Number analyzed (Participants) | 155
percentage of subjects | 59.4

6. Secondary Outcome: Percentage of Subjects With ACR70 (American College of Rheumatology 70% Improvement) Response at Completion/Withdrawal Visit
Description: ACR70 response is defined for subjects with at least 70% improvement from Baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: 1) Health Assessment Questionnaire-Disability Index (HAQ-DI), 2) C-reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale, 4) Patient's Global Assessment of Disease Activity, 5) Physician's Global Assessment of Disease Activity.
Time Frame: Baseline (in C87077 [NCT00580840]) to Completion/Withdrawal Visit (up to approximately 54 weeks)
Population: as for outcome 4
Measure: Number; unit: percentage of subjects
Arm/Group | CDP870
Number analyzed (Participants) | 155
percentage of subjects | 39.4

7. Secondary Outcome: Change From Baseline in DAS28[ESR] (Disease Activity Score 28 [Erythrocyte Sedimentation Rate]) at Completion/Withdrawal Visit
Description: DAS28(ESR) is calculated using the tender joint count (TJC), swollen joint count (SJC) erythrocyte sedimentation rate (ESR in mm/hour), and the Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS in mm) using the following formula: 0.56 x √(TJC) + 0.28 x √(SJC) + 0.70 x lognat (ESR) + 0.014 x Global Assessment of Arthritis where 28 joints are examined and a lower score indicates less disease activity. This analysis was carried out using the Last Observation Carried Forward (LOCF) method.
  < 2.6 Remission,
  > = 2.6 - < =3.2 Low, > 3.2 - < = 5.1 Moderate, > 5.1 High.
Time Frame: Baseline (in C87077 [NCT00580840]) to Completion/Withdrawal Visit (up to approximately 54 weeks)
Population: Of the 168 subjects in the Full Analysis Set (FAS), 142 are included in this analysis.
  Data was not available for 26 subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CDP870
Number analyzed (Participants) | 142
units on a scale | -2.94 (1.33)

8. Secondary Outcome: Change From Baseline in SDAI (Simplified Disease Activity Index) at Completion/Withdrawal Visit
Description: SDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), C-reactive protein (CRP in mg/dL), Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS in cm), and Investigator's Global Assessment of Disease Activity - Visual Analog Scale (VAS in cm). 28 joints are examined where a lower score indicates less disease activity. This analysis was carried out using the Last Observation Carried Forward (LOCF) method.
  <= 3.3 Remission, > 3.3 - <= 11 Low, > 11 - <= 26 Moderate, > 26 High.
Time Frame: Baseline (in C87077 [NCT00580840]) to Completion/Withdrawal Visit (up to approximately 54 weeks)
Population: Of the 168 subjects in the Full Analysis Set (FAS), 145 are included in this analysis.
  Data was not available for 23 subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CDP870
Number analyzed (Participants) | 145
units on a scale | -29.14 (14.62)

9. Secondary Outcome: Change From Baseline in CDAI (Clinical Disease Activity Index) at Completion/Withdrawal Visit
Description: CDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS in cm), and Investigator's Global Assessment of Disease Activity - Visual Analog Scale (VAS in cm). 28 joints are examined. This analysis was carried out using the Last Observation Carried Forward (LOCF) method.
  The range for the CDAI is 0 - 76 with a negative change in CDAI score indicating an improvement in disease activity and a positive change in score indicating a worsening of disease activity.
Time Frame: Baseline (in C87077 [NCT00580840]) to Completion/Withdrawal Visit (up to approximately 54 weeks)
Population: Of the 168 subjects in the Full Analysis Set (FAS), 146 are included in this analysis.
  Data was not available for 22 subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CDP870
Number analyzed (Participants) | 146
units on a scale | -28.26 (13.94)

10. Secondary Outcome: Percentage of Subjects With DAS28[ESR] (Disease Activity Score 28 [Erythrocyte Sedimentation Rate]) Remission (DAS28[ESR] < 2.6) at Completion/Withdrawal Visit
Description: DAS28(ESR) is calculated using the tender joint count (TJC), swollen joint count (SJC) erythrocyte sedimentation rate (ESR in mm/hour), and the Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS in mm) using the following formula: 0.56 x √(TJC) + 0.28 x √(SJC) + 0.70 x lognat (ESR) + 0.014 x Global Assessment of Arthritis where 28 joints are examined and a lower score indicates less disease activity. Missing values were imputed using Non-Responder Imputation (NRI).
  < 2.6 (Remission),
  > = 2.6 - < =3.2 Low, > 3.2 - < = 5.1 Moderate, > 5.1 High.
Time Frame: Baseline (in C87077 [NCT00580840]) to Completion/Withdrawal Visit (up to approximately 54 weeks)
Population: Of the 168 subjects in the Full Analysis Set (FAS), 149 are included in this analysis.
  Data was not available for 19 subjects.
Measure: Number; unit: percentage of subjects
Arm/Group | CDP870
Number analyzed (Participants) | 149
percentage of subjects | 32.9

11. Secondary Outcome: Percentage of Subjects With SDAI (Simplified Disease Activity Index) Remission (SDAI ≤3.3) at Completion/Withdrawal Visit
Description: SDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), C-reactive protein (CRP in mg/dL), Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS in cm), and Investigator's Global Assessment of Disease Activity - Visual Analog Scale (VAS in cm). 28 joints are examined where a lower score indicates less disease activity. Missing values were imputed using Non-Responder Imputation (NRI).
  <= 3.3 (Remission), > 3.3 - <= 11 Low, > 11 - <= 26 Moderate, > 26 High.
Time Frame: Baseline (in C87077 [NCT00580840]) to Completion/Withdrawal Visit (up to approximately 54 weeks)
Population: Of the 168 subjects in the Full Analysis Set (FAS), 151 are included in this analysis.
  Data was not available for 17 subjects.
Measure: Number; unit: percentage of subjects
Arm/Group | CDP870
Number analyzed (Participants) | 151
percentage of subjects | 31.1

12. Secondary Outcome: Percentage of Subjects With CDAI (Clinical Disease Activity Index) Remission (CDAI ≤2.8) at Completion/Withdrawal Visit
Description: CDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS in cm), and Investigator's Global Assessment of Disease Activity - Visual Analog Scale (VAS in cm). 28 joints are examined where a lower score indicates less disease activity. Missing values were imputed using Non-Responder Imputation (NRI).
  The range for the CDAI is 0 - 76 with a lower CDAI score indicating improvement in activity and a higher score indicating a decline activity.
Time Frame: Baseline (in C87077 [NCT00580840]) to Completion/Withdrawal Visit (up to approximately 54 weeks)
Population: Of the 168 subjects in the Full Analysis Set (FAS), 152 are included in this analysis.
  Data was not available for 16 subjects.
Measure: Number; unit: percentage of subjects
Arm/Group | CDP870
Number analyzed (Participants) | 152
percentage of subjects | 30.3

13. Secondary Outcome: Change From Baseline in HAQ-DI (Health Assessment Questionnaire-Disability Index) at Completion/Withdrawal Visit
Description: HAQ-DI is derived based on the mean of individual scores in 8 categories of daily living actives (using 20 questions). Each question is scored 0-3 (0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do). Thus, the mean also has a range from 0-3. Change from Baseline is computed as the value at Completion/Withdrawal minus the Baseline value. A negative value in change from Baseline indicates an improvement. This analysis was carried out using the Last Observation Carried Forward (LOCF) method.
Time Frame: Baseline (in C87077 [NCT00580840]) to Completion/Withdrawal Visit (up to approximately 54 weeks)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CDP870
Number analyzed (Participants) | 142
units on a scale | -0.67 (0.59)

14. Secondary Outcome: Change From Baseline in FAS (Fatigue Assessment Scale) at Completion/Withdrawal Visit
Description: Change from Baseline in Fatigue Assessment scale (0 to 10, 0 is "No Fatigue" and 10 is "Fatigue as bad as you can imagine") is computed as the value at Completion/Withdrawal minus the Baseline value. A negative value in change from Baseline indicates an improvement. This analysis was carried out using the Last Observation Carried Forward (LOCF) method.
Time Frame: Baseline (in C87077 [NCT00580840]) to Completion/Withdrawal Visit (up to approximately 54 weeks)
Population: Of the 168 subjects in the Full Analysis Set (FAS), 139 are included in this analysis.
  Data was not available for 29 subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CDP870
Number analyzed (Participants) | 139
units on a scale | -2.58 (2.51)

15. Secondary Outcome: Change From Baseline in Physical Functioning (Short Form 36-item Health Survey Domain) at Completion/Withdrawal Visit
Description: There are 8 SF-36 domain scores: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional and Mental Health, each ranging from 0 to 100, with higher scores indicating better health. A larger positive value in change from Baseline indicates an improvement. This analysis was carried out using the Last Observation Carried Forward (LOCF) method.
Time Frame: Baseline (in C87077 [NCT00580840]) to Completion/Withdrawal Visit (up to approximately 54 weeks)
Population: Of the 168 subjects in the Full Analysis Set (FAS), 143 are included in this analysis.
  Data was not available for 25 subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CDP870
Number analyzed (Participants) | 143
units on a scale | 9.04 (9.69)

16. Secondary Outcome: Change From Baseline in Role Physical (Short Form 36-item Health Survey Domain) at Completion/Withdrawal Visit
Description: as for outcome 15
Time Frame: Baseline (in C87077 [NCT00580840]) to Completion/Withdrawal Visit (up to approximately 54 weeks)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CDP870
Number analyzed (Participants) | 143
units on a scale | 10.32 (10.5)

17. Secondary Outcome: Change From Baseline in Bodily Pain (Short Form 36-item Health Survey Domain) at Completion/Withdrawal Visit
Description: as for outcome 15
Time Frame: Baseline (in C87077 [NCT00580840]) to Completion/Withdrawal Visit (up to approximately 54 weeks)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CDP870
Number analyzed (Participants) | 143
units on a scale | 12.73 (8.9)

18. Secondary Outcome: Change From Baseline in General Health (Short Form 36-item Health Survey Domain) at Completion/Withdrawal Visit
Description: as for outcome 15
Time Frame: Baseline (in C87077 [NCT00580840]) to Completion/Withdrawal Visit (up to approximately 54 weeks)
Population: Of the 168 subjects in the Full Analysis Set (FAS), 141 are included in this analysis.
  Data was not available for 27 subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CDP870
Number analyzed (Participants) | 141
units on a scale | 5.1 (7.9)

19. Secondary Outcome: Change From Baseline in Vitality (Short Form 36-item Health Survey Domain) at Completion/Withdrawal Visit
Description: as for outcome 15
Time Frame: Baseline (in C87077 [NCT00580840]) to Completion/Withdrawal Visit (up to approximately 54 weeks)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CDP870
Number analyzed (Participants) | 141
units on a scale | 10.27 (10.27)

20. Secondary Outcome: Change From Baseline in Social Functioning (Short Form 36-item Health Survey Domain) at Completion/Withdrawal Visit
Description: as for outcome 15
Time Frame: Baseline (in C87077 [NCT00580840]) to Completion/Withdrawal Visit (up to approximately 54 weeks)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CDP870
Number analyzed (Participants) | 143
units on a scale | 8.54 (12.29)

21. Secondary Outcome: Change From Baseline in Role Emotional (Short Form 36-item Health Survey Domain) at Completion/Withdrawal Visit
Description: as for outcome 15
Time Frame: Baseline (in C87077 [NCT00580840]) to Completion/Withdrawal Visit (up to approximately 54 weeks)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CDP870
Number analyzed (Participants) | 141
units on a scale | 7 (13.56)

22. Secondary Outcome: Change From Baseline in Mental Health (Short Form 36-item Health Survey Domain) at Completion/Withdrawal Visit
Description: as for outcome 15
Time Frame: Baseline (in C87077 [NCT00580840]) to Completion/Withdrawal Visit (up to approximately 54 weeks)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CDP870
Number analyzed (Participants) | 141
units on a scale | 5.57 (9.55)

23. Secondary Outcome: Change From Baseline in PCS (Short Form 36-item Health Survey Physical Component Summary) at Completion/Withdrawal Visit
Description: PCS norm-based scores are calculated based upon the following 8 domain scores, Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional and Mental Health, and range from 1 to 81, where 50 represents the normative value. A larger positive value in change from Baseline indicates an improvement. This analysis was carried out using the Last Observation Carried Forward (LOCF) method.
Time Frame: Baseline (in C87077 [NCT00580840]) to Completion/Withdrawal Visit (up to approximately 54 weeks)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CDP870
Number analyzed (Participants) | 139
units on a scale | 10.73 (8.56)

24. Secondary Outcome: Change From Baseline in MCS (Short Form 36-item Health Survey Mental Component Summary) at Completion/Withdrawal Visit
Description: MCS norm-based scores are calculated based upon the following 8 domain scores, Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional and Mental Health, and range from -9 to 82, where 50 represents the normative value. A larger positive value in change from Baseline indicates an improvement. This analysis was carried out using the Last Observation Carried Forward (LOCF) method.
Time Frame: Baseline (in C87077 [NCT00580840]) to Completion/Withdrawal Visit (up to approximately 54 weeks)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CDP870
Number analyzed (Participants) | 139
units on a scale | 5.82 (11.3)

25. Secondary Outcome: Change From Baseline in PtAAP (Patient's Assessment of Arthritis Pain) at Completion/Withdrawal Visit
Description: Change from Baseline in Patient's Assessment of Arthritis Pain-VAS (0 to 100 mm visual analog scale, 0 being no pain and 100 being most severe pain) is computed as the value at Completion/Withdrawal minus the Baseline value. A negative value in change from Baseline indicates an improvement. This analysis was carried out using the Last Observation Carried Forward (LOCF) method.
Time Frame: Baseline (in C87077 [NCT00580840]) to Completion/Withdrawal Visit (up to approximately 54 weeks)
Population: Of the 168 subjects in the Full Analysis Set (FAS), 140 are included in this analysis.
  Data was not available for 28 subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CDP870
Number analyzed (Participants) | 140
units on a scale | -36.04 (27.72)

26. Secondary Outcome: Change From Baseline in PtGADA (Patient's Global Assessment of Disease Activity) at Completion/Withdrawal Visit
Description: Change from Baseline in Patient's Global Assessment of Disease Activity-VAS (0 to 100 mm visual analog scale, 0 being no symptoms and 100 being severe symptoms) is computed as the value at Completion/Withdrawal minus the Baseline value. A negative value in change from Baseline indicates an improvement. This analysis was carried out using the Last Observation Carried Forward (LOCF) method.
Time Frame: Baseline (in C87077 [NCT00580840]) to Completion/Withdrawal Visit (up to approximately 54 weeks)
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CDP870
Number analyzed (Participants) | 140
units on a scale | -35.51 (27.49)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from Entry Visit up to approximately 60 weeks.
Description: Adverse Events refer to the Safety Set (SS). SS includes all subjects that were administered the investigational product at least once.
Arm/Group | CDP870
Serious Adverse Events (participants affected / at risk) | 5/168
Other Adverse Events (participants affected / at risk) | 23/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CDP870 (N=168)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Perirectal Abscess (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neuropathy Peripheral (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CDP870 (N=168)
Upper Respiratory Tract Infection (Infections and infestations) | 23 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that the results shall be published regardless of outcome.